CLINICAL TRIAL: NCT04255095
Title: Application of Negative Pressure Suction in Nasopancreatic Duct in Patients With Severe Biliary Pancreatitis
Brief Title: Early Intervention of High Tension in the Pancreatic Duct on the Outcome of Severe Biliary Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERCP-0001
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: ERCP
Keywords: Pancreatic duct negative-pressure suction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasobiliary drainage (Active Comparator)
  Interventions: Procedure: control
- Naso-pancreatic drainage(negative pressure) (Experimental)
  Interventions: Procedure: experiment

INTERVENTIONS:
Procedure: experiment — Treatment was randomly selected according to preoperative grouping. After ERCP, naso-pancreatic drainage was chosen as treatment。
  Other Names: Naso-pancreatic duct negative pressure attraction
  Arms: Naso-pancreatic drainage(negative pressure)
Procedure: control — Treatment was randomly selected according to preoperative grouping. After ERCP, nasobiliary drainage was chosen as treatment。
  Other Names: naso-biliary drinage
  Arms: Nasobiliary drainage

SUMMARY:
The investigators hypothesized that naso-pancreatic duct suction could benefit for patients with severe biliary pancreatitis undergoing ERCP. So, the investigators designed this experiment to verify it.

DETAILED DESCRIPTION:
This project intends to conduct treatment based on different interventions for enrolled subjects according to international and domestic standardized treatment procedures, including 1.ERCP stone extraction, duodenal papillary pressure measurement, bile duct pressure measurement, and nasal bile duct placement; 2.ERCP+ duodenal papillary pressure measurement, biliopancreatic duct pressure measurement + nasopancreatic duct + determine whether nasopancreatic duct negative pressure attraction.Compare the advantages of two different treatment methods.This paper attempts to explore new treatment methods that are more conducive to the rehabilitation of patients and provides an important preliminary research basis for the future clinical application of standardized treatment.

Patients from the people's hospital of Wuhan university were recruited and selected into groups. The incidence, recurrence rate, operation time and hospital stay of the two independent samples will be compared.

ELIGIBILITY:
Inclusion Criteria:

Ages 16 to 75. Apach-ii score of patients diagnosed with pancreatitis was greater than 8 points.

Liver function can be damaged. Elevated indicators of pancreatitis (hematuria amylase, lipase). Identify patients with biliary tract infection or obstruction.

Exclusion Criteria:

Older than 75 or younger than 16. The duration of admission was more than 72 hours. Gastrointestinal obstruction endoscopy cannot be operated. Patients with duodenoscopy contraindications.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Rehabilitation | 2 months
  time from ERCP to ischarge
complication rate | 1 months
  Pancreatitis aggravation， hemorrhage，fistula

SECONDARY OUTCOMES:
LOS(length of stay) | postoperative period（1 month ）
  time from operation to discharge
death rate | postoperative period（1 month ）
  Mortality from the disease

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China